CLINICAL TRIAL: NCT00508547
Title: A Multicenter, Open Registry of Patients With Plaque Psoriasis Who Are Candidates for Systemic Therapy Including Biologics
Brief Title: Psoriasis Longitudinal Assessment and Registry
Acronym: PSOLAR
Status: Active, not recruiting | Type: Observational
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR013225; C0168Z03 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis
Keywords: psoriasis; psoriatic arthritis; skin disease; infliximab; ustekinumab; guselkumab; etanercept; adalimumab; secukinumab; ixekizumab; brodalumab; systemic therapy; observational; registry
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic; Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Guselkumab: Participants will receive guselkumab as prescribed by a physician according to standard of care for psoriasis.
- Infliximab: Participants will receive infliximab as prescribed by a physician according to standard of care for psoriasis.
- Ustekinumab: Participants will receive ustekinumab as prescribed by a physician according to standard of care for psoriasis.
- Biological Therapies: Participants will receive biological therapies other than infliximab, ustekinumab, guselkumab, and IL-17 inhibitors as prescribed by a physician for psoriasis. Participants will not receive any intervention as a part of this study.
- Conventional Systemic Agents: Participants will receive conventional systemic agents as prescribed by a physician for psoriasis. Participants will not receive any intervention as a part of this study.
- IL-17 Inhibitor: Participants will receive an IL-17 inhibitor as prescribed by a physician according to standard of care for psoriasis.

SUMMARY:
The purpose of this study is to further evaluate the safety of infliximab, ustekinumab, and guselkumab in patients with plaque and other forms of psoriasis. The study also includes patients receiving other therapies, such as non-biologic and other biologic agents. The registry also evaluates patient and disease characteristics, including patient-reported assessment of psoriatic arthritis (PsA); and clinical and quality of life outcomes.

DETAILED DESCRIPTION:
PSOLAR is an ongoing voluntary observational study in which infliximab-exposed patients, ustekinumab-exposed patients, and patients treated with other biologic and non-biologic standard of care therapies have been enrolled internationally and are followed for up to 8 years. Additionally, enrollment is opened to include at least 2000 guselkumab-exposed patients and up to 2000 patients exposed to IL-17 inhibitors. The Registry does not require any study-specific testing, but may capture information collected as part of normal routine care. Patient information is collected at the enrollment visit and about every 6 months thereafter. At enrollment, information on demographics (e.g. gender, and race), medical history and family medical history, details of past and current psoriasis treatments, and current psoriasis medications is collected. At enrollment and each follow-up visit, data are collected regarding physical examination, clinical disease status, Quality of Life assessments, current psoriasis medications, patient-reported PsA assessments, and adverse events. No study agents are administered for the purpose of this registry; all patients receive standard of care treatment as prescribed by the patient's physician.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of psoriasis
* Incident or prevalent users of Tremfya or an IL-17 inhibitor (eg, secukinumab, ixekizumab, brodalumab, bimekizumab) at the time of their enrollment. Incident users are defined as those participants starting treatment within 30 days before or after the enrollment visit and prevalent users are defined as those who are on treatment greater than 30 days prior to the enrollment visit
* Ability to understand and sign an informed consent form
* Are willing to participate in regular follow-up visits

Exclusion Criteria:

* Refuse to consent or are unwilling to respond to requests for long term information within the required time frame
* Are participating or have already planned to participate in a clinical trial with non-marketed investigational agents or are participating in a Janssen-sponsored clinical trial with marketed agents

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with psoriasis who meets the inclusion criteria will be eligible to participate in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 15842 (Actual)
Dates: Start 2007-06-21 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events and Serious Adverse Events | Up to 8 years of follow up for each patient
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; suspected transmission of any infectious agent via medicinal product; any important medical events. All adverse events, including those of special interest, such as malignancies;TB;opportunistic infections;depression;hypersensitivity reactions; autoimmune disease; neurologic or demyelinating events; congestive heart failure; gastrointestinal events; demyelinating disease, hepatotoxicity; hematologic events; unexpected reaction to a vaccine;cerebrovascular accident; transient ischemic attack; confirmed myocardial infarction; acquired immunodeficiency syndrome will be documented.

SECONDARY OUTCOMES:
Evaluation of disease features: Physicians global assessment of disease activity (PGA) Score | At baseline and every 6 months through up to 8 years
Evaluation of Disease Features: Body surface area | At baseline and every 6 months through up to 8 years
Evaluation of Disease Features: Psoriasis Area and Severity Index (PASI) Score | At baseline and every 6 months through up to 8 years
Dermatology Life Quality Index (DLQI) Score | At baseline and every 6 months through up to 8 years
EuroQOL quality of life assessment | At baseline and every 6 months through up to 8 years
Hospital Anxiety and Depression Scale (HADS) Score | At baseline and every 6 months up to Month 18 and then every year up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (319):
- United States (167):
  - Birmingham, Alabama
  - Florence, Alabama
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Rogers, Arkansas
  - Bakersfield, California
  - Clovis, California
  - Fountain Valley, California
  - Fresno, California
  - Loma Linda, California
  - Los Angeles, California
  - Mountain View, California
  - Oxnard, California
  - Redding, California
  - Rolling Hills Estates, California
  - San Diego, California
  - San Ramon, California
  - Santa Monica, California
  - Sherman Oaks, California
  - Upland, California
  - Vallejo, California
  - Colorado Springs, Colorado
  - Englewood, Colorado
  - Bridgeport, Connecticut
  - Farmington, Connecticut
  - Newark, Delaware
  - Wilmington, Delaware
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Bay Pines, Florida
  - Boca Raton, Florida
  - Boynton Beach, Florida
  - Coral Gables, Florida
  - Delray Beach, Florida
  - Dunedin, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Naples, Florida
  - North Miami Beach, Florida
  - Panama City, Florida
  - Pembroke Pines, Florida
  - Seminole, Florida
  - Tampa, Florida
  - Alpharetta, Georgia
  - Atlanta, Georgia
  - Birmingham, Georgia
  - Carrollton, Georgia
  - Conyers, Georgia
  - Lilburn, Georgia
  - Macon, Georgia
  - Marietta, Georgia
  - Rome, Georgia
  - Twin Falls, Idaho
  - Champaign, Illinois
  - Chicago, Illinois
  - Lincolnshire, Illinois
  - Maywood, Illinois
  - Rolling Meadows, Illinois
  - Schaumburg, Illinois
  - Skokie, Illinois
  - Springfield, Illinois
  - West Dundee, Illinois
  - Winfield, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - New Albany, Indiana
  - Plainfield, Indiana
  - West Lafayette, Indiana
  - Topeka, Kansas
  - Corbin, Kentucky
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Quincy, Massachusetts
  - Ann Arbor, Michigan
  - Clarkston, Michigan
  - Clinton Township, Michigan
  - Farmington, Michigan
  - Flint, Michigan
  - Fort Gratiot, Michigan
  - Grand Blanc, Michigan
  - Grand Rapids, Michigan
  - Monroe, Michigan
  - Norton Shores, Michigan
  - Troy, Michigan
  - Warren, Michigan
  - Eagan, Minnesota
  - Chesterfield, Missouri
  - St Louis, Missouri
  - Helena, Montana
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Nashua, New Hampshire
  - Belleville, New Jersey
  - East Windsor, New Jersey
  - Hoboken, New Jersey
  - Marlton, New Jersey
  - Rutherford, New Jersey
  - Somerset, New Jersey
  - Verona, New Jersey
  - Wyckoff, New Jersey
  - Auburn, New York
  - Commack, New York
  - East Syracuse, New York
  - Elmhurst, New York
  - Garden City, New York
  - Huntington, New York
  - Lawrence, New York
  - New York, New York
  - Oceanside, New York
  - Rochester, New York
  - Smithtown, New York
  - Staten Island, New York
  - Stony Brook, New York
  - Suffern, New York
  - Syracuse, New York
  - The Bronx, New York
  - White Plains, New York
  - Williamsville, New York
  - Chapel Hill, North Carolina
  - Raleigh, North Carolina
  - Rocky Mount, North Carolina
  - Wilmington, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Delaware, Ohio
  - Gahanna, Ohio
  - Warren, Ohio
  - Oklahoma City, Oklahoma
  - Coos Bay, Oregon
  - Portland, Oregon
  - Exton, Pennsylvania
  - Fort Washington, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Plymouth Meeting, Pennsylvania
  - Charleston, South Carolina
  - Fort Mill, South Carolina
  - Piedmont, South Carolina
  - Spartanburg, South Carolina
  - Bartlett, Tennessee
  - Bristol, Tennessee
  - Kingsport, Tennessee
  - Arlington, Texas
  - Cedar Hill, Texas
  - Dallas, Texas
  - Houston, Texas
  - Longview, Texas
  - Salt Lake City, Utah
  - Arlington, Virginia
  - Norfolk, Virginia
  - Kennewick, Washington
  - Mount Vernon, Washington
  - Seattle, Washington
  - Tacoma, Washington
  - University Place, Washington
  - Walla Walla, Washington
  - Green Bay, Wisconsin
  - Pleasant Prairie, Wisconsin
  - Sheboygan, Wisconsin
- Argentina (5):
  - Buenos Aires
  - CABA
  - Cipolletti
  - Lomas de Zamora
  - San Miguel
- Australia (5):
  - Fremantle
  - Melbourne
  - Miranda
  - Sydney
  - Woolloongabba
- Austria (8):
  - Althofen
  - Feldkirch
  - Graz
  - Klagenfurt
  - Laakirchen
  - Sankt Pölten
  - Vienna
  - Villach
- Belgium (7):
  - Bruges
  - Brussels
  - Edegem
  - Ghent
  - Leuven
  - Liège
  - Mons
- Canada (30):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Nanaimo, British Columbia
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Fredericton, New Brunswick
  - Moncton, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Kentville, Nova Scotia
  - Barrie, Ontario
  - Coburg, Ontario
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Kingston, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Markham, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - North Bay, Ontario
  - Ottawa, Ontario
  - Peterborough, Ontario
  - Saint Catherines, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Drummondville, Quebec
  - Montreal, Quebec
  - Québec, Quebec
- Chile (3):
  - Santiago
  - Santiago - Las Condes
  - Santiago - Macul
- Colombia (2):
  - Bogotá
  - Medellín
- Czechia (11):
  - Brno
  - České Budějovice
  - Jihlava
  - Náchod
  - Nový Jičín
  - Olomouc
  - Pardubice
  - Pilsen
  - Prague
  - Šumperk
  - Ústí nad Labem
- Greece (7):
  - Athens
  - Heraklion
  - Ioannina
  - Larissa
  - Pátrai
  - Piraeus-Athens
  - Thessaloniki
- Israel (7):
  - Afula
  - Beersheba
  - Haifa
  - Netivot
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Japan (11):
  - Hirakata
  - Hokkaido
  - Itabashi Ku
  - Kobe
  - Kurume
  - Matsumoto
  - Ōita
  - Takamatsu
  - Tokyo
  - Tsu
  - Yokosuka
- Mexico (4):
  - Estado de México
  - Mexico City
  - Monterrey
  - Zapopan
- Netherlands (6):
  - Alkmaar
  - Amsterdam-Zuidoost
  - Breda
  - Deventer
  - Helmond
  - Nijmegen
- Portugal (4):
  - Braga
  - Lisbon
  - Porto
  - Vila Nova de Gaia
- Slovakia (8):
  - Banská Bystrica
  - Bratislava
  - Košice
  - Martin
  - Nitra
  - Poprad
  - Prešov
  - Trnava
- Slovenia (5):
  - Celje
  - Izola
  - Kranj
  - Ljubljana
  - Maribor
- South Korea (5):
  - Busan
  - Gyeonggi-do
  - Seongnam-si
  - Seoul
  - Sungnam
- Spain (8):
  - Alcalá de Henares
  - Bilbao
  - Granada
  - Madrid
  - Majadahonda
  - Murcia
  - Salamanca
  - Santiago de Compostela
- Sweden (4):
  - Eskilstuna
  - Gothenburg
  - Kungsbacka
  - Stockholm
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan
- Ukraine (8):
  - Dnipro
  - Donetsk
  - Kharkiv
  - Khmelnitskiy
  - Kiev
  - Luhansk
  - Simferopol
  - Uzhhorod

REFERENCES:
- [Derived] Ritchlin CT, Stahle M, Poulin Y, Bagel J, Chakravarty SD, Kafka S, Srivastava B, Langholff W, Gottlieb AB. Serious infections in patients with self-reported psoriatic arthritis from the Psoriasis Longitudinal Assessment and Registry (PSOLAR) treated with biologics. BMC Rheumatol. 2019 Nov 28;3:52. doi: 10.1186/s41927-019-0094-3. eCollection 2019. PMID 31799498
- [Derived] Kavanaugh A, Papp K, Gottlieb AB, de Jong EMGJ, Chakravarty SD, Kafka S, Langholff W, Farahi K, Srivastava B, Scher JU. Demography, baseline disease characteristics, and treatment history of psoriasis patients with self-reported psoriatic arthritis enrolled in the PSOLAR registry. BMC Rheumatol. 2018 Sep 29;2:29. doi: 10.1186/s41927-018-0034-7. eCollection 2018. PMID 30886979
- [Derived] Singh S, Kalb RE, de Jong EMGJ, Shear NH, Lebwohl M, Langholff W, Hopkins L, Srivastava B, Armstrong AW. Effect of Age of Onset of Psoriasis on Clinical Outcomes with Systemic Treatment in the Psoriasis Longitudinal Assessment and Registry (PSOLAR). Am J Clin Dermatol. 2018 Dec;19(6):879-886. doi: 10.1007/s40257-018-0388-z. PMID 30267377
- [Derived] Strober BE, Bissonnette R, Fiorentino D, Kimball AB, Naldi L, Shear NH, Goyal K, Fakharzadeh S, Calabro S, Langholff W, You Y, Galindo C, Lee S, Lebwohl MG. Comparative effectiveness of biologic agents for the treatment of psoriasis in a real-world setting: Results from a large, prospective, observational study (Psoriasis Longitudinal Assessment and Registry [PSOLAR]). J Am Acad Dermatol. 2016 May;74(5):851-61.e4. doi: 10.1016/j.jaad.2015.12.017. Epub 2016 Feb 4. PMID 26853180
- [Derived] Kalb RE, Fiorentino DF, Lebwohl MG, Toole J, Poulin Y, Cohen AD, Goyal K, Fakharzadeh S, Calabro S, Chevrier M, Langholff W, You Y, Leonardi CL. Risk of Serious Infection With Biologic and Systemic Treatment of Psoriasis: Results From the Psoriasis Longitudinal Assessment and Registry (PSOLAR). JAMA Dermatol. 2015 Sep;151(9):961-9. doi: 10.1001/jamadermatol.2015.0718. PMID 25970800